CLINICAL TRIAL: NCT06665724
Title: A Phase 1 Single Center Clinical Trial Evaluating Safety of 5-Aminolevulinic Acid (5-ALA) Combined With CV01 Delivery of Ultrasound for Sonodynamic Therapy (SDT) in Patients With Newly Diagnosed High-Grade Glioma (HGG) Prior to Resection and Standard Adjuvant Therapy
Brief Title: Clinical Trial Evaluating Safety of 5-Aminolevulinic Acid (5-ALA) Combined With CV01 Delivery of Ultrasound for Sonodynamic Therapy (SDT) in Patients With Newly Diagnosed High-Grade Glioma (HGG) Prior to Resection and Standard Adjuvant Therapy (ALA SDT GLIOMA 401)
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Universität Münster (Other)
Collaborators: Alpheus Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WWU22_0032; 2023-509238-20-00 (EU CTIS Number); UTN: U1111-1296-1261 (Other: WHO)
Record Dates: First submitted 2024-10-29; First posted 2024-10-30 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Anaplastic Astrocytoma (AA); Anaplastic Oligodendroglioma (AO); Glioblastoma (GBM)
Keywords: newly diagnosed high-grade glioma; sonodynamic therapy
MeSH Terms: conditions — Astrocytoma; Oligodendroglioma; Glioblastoma | interventions — Aminolevulinic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sonodynamic Therapy (SDT) (Experimental): Patients will receive sonodynamic therapy (5 ALA combined with CV01-delivered sonication) 2 to 5 days prior to standard resection.
  Interventions: Drug: 5-Aminolevulinic acid Hydrochloride (Gliolan®); Device: CV01

INTERVENTIONS:
Drug: 5-Aminolevulinic acid Hydrochloride (Gliolan®) — Patients will receive 5-Aminolevulinic acid hydrochloride via oral administration (20 mg/kg) 6-8 hours before CV01 treatment.
Device: CV01 — Ultrasound will be delivered 6-8 hours after administration of 5-aminolevulinic acid hydrochloride. A total of 12 fields will be treated (10 treatment sites across the hemisphere with 2 additional treatments over areas of increased enhancement).

SUMMARY:
This trial is designed to evaluate safety and explore possible efficacy of 5-aminolevulinic acid hydrochloride (5-ALA HCl, Gliolan®) with CV01 delivery of ultrasound for sonodynamic therapy in patients with newly diagnosed high-grade glioma prior to resection and standard adjuvant therapy.

The study will accrue 10 evaluable high-grade glioma patients. Patients who qualify will receive sonodynamic therapy (5 ALA combined with CV01-delivered sonication) 2 to 5 days prior to standard resection, with one study magnetic resonance imaging being performed between sonodynamic therapy and resection. Resection will be followed by standard radio-/chemotherapy. All patients will be followed up in-study for toxicities and adverse events for 28 days.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. WHO Performance Status of 0-2
3. Patients with cranial MRI displaying typical features of high-grade glioma on imaging or histologically proven high-grade glioma including GBM, anaplastic astrocytoma (AA), anaplastic oligodendroglioma (AO). No previous tumor specific treatment such as surgery (apart from biopsy), radio- or chemotherapy, antiangiogenic or immunotherapy.
4. Planned debulking or cytoreductive surgery
5. The following laboratory values at study entry

   1. Absolute neutrophil count (ANC) ≥ 1500 cells/mm3
   2. Platelet count ≥ 100,000 cells/mm3
   3. Hemoglobin (Hgb) > 10g/dL
   4. AST and ALT ≤ 2.5 x Upper Limit of Normal (ULN)
   5. Total bilirubin ≤ 1.5 x ULN
   6. Creatine clearance (CrCL) as estimated by Cockcroft-Gault equation of

      ≥ 40 mL/min
   7. Blood clotting within acceptable limits according to investigator
6. For female and male patients and their female partners of childbearing/reproductive potential: Willingness to apply highly effective contraception (Pearl index <1) during the entire study and in female patients for 6 months after the last application of Gliolan® and in male patients and their female partners for 3 months after the last application of Gliolan®.
7. Ability to understand and provide informed consent

Exclusion Criteria:

1. Infra-tentorial tumors
2. Patients who have clinically significant edema or tumor mass effect requiring urgent intervention (e.g., surgery, initiation of steroids, escalating doses of steroids)
3. Women who are pregnant or breastfeeding
4. Inability to undergo MRI or receive gadolinium (Gd)
5. Hypersensitivity to 5-ALA or porphyrins
6. Average skull thickness at the treatment field > 10 mm from standard navigation CTs. The treatment field is defined as the various locations on the head where the transducer will be coupled to the patient. The average skull thickness at each treatment field will be determined through post-processing the thin cut head computed tomography (CT) scan (without contrast).
7. Hemorrhagic or ischemic stroke (including transient ischemic attacks) and central nervous system bleeding in the preceding 6 months that are not related to glioma biopsy. History of prior intratumoral bleeding is not an exclusion criterion; however, all patient's navigation CTs will be reviewed for the presence of fresh blood.
8. Participation in another interventional clinical trial during this trial or within 4 weeks before entry into this trial
9. Known acute or chronic types of porphyria
10. Gastrointestinal disorder that negatively affects absorption
11. Known active hepatitis B or C (Note: testing is not required)
12. Known Human Immunodeficiency Virus (HIV) infection (Note: testing is not required)
13. Unable to avoid photosensitising drugs (eg, St. John's wort, griseofulvin, thiazide diuretics, sulfonylureas, phenothiazines, sulfonamides, quinolones, and tetracyclines) for up to 2 weeks following 5-ALA administration
14. Any other concurrent severe and/or uncontrolled concomitant medical condition that could compromise participation in the study (e.g, clinically significant pulmonary disease, clinically significant psychiatric or neurological disorder, active or uncontrolled infection)
15. Diagnosis of other invasive cancer (except basal cell carcinoma/squamous cell carcinoma of the skin) within the last 5 years; adequately treated carcinoma in situ is allowed
16. Patient has a condition the investigator believes would interfere with the ability to provide informed consent or comply with study instructions, or that might confound the interpretation of the study results or put the patient at undue risk
17. Patients who are dependent on the sponsor, investigator or trial site
18. Patients who are committed to an institution by virtue of an order issued either by the judicial or the administrative authorities

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Estimated)
Dates: Start 2025-01-27 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability | From the time the informed consent is signed until 28 days following administration of sonodynamic therapy (end of trial participation)
  Clinical safety and tolerability will be assessed based on the observation of adverse events (AEs). Adverse events will be graded as per the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) v5.

SECONDARY OUTCOMES:
Radiological changes | Changes from visit 1 (< 8 days before sonodynamic therapy) to visit 3 (2 to 5 days after sonodynamic therapy)
  Radiological changes (MRI) of Tumor volume, Volume of FLAIR hyperintensity, Volume of cyctotoxic edema, Relative cerebral blood volume and Leakage
Histopathological efficacy | Biopsies will be collected during standard surgery.
  Anti-tumor activity assessed by Number of cells / mm³ with antibodies against IBA1 and Number of cells / mm³ with antibodies against Caspase III

CONTACTS AND LOCATIONS:
Overall Officials: Walter Stummer, Univ.-Prof. Dr. med., Principal Investigator — Department of Neurosurgery, University Hospital Münster, Münster, Germany, 48149
Locations (1):
- Department of Neurosurgery, University Hospital Münster, Münster, Germany

IPD SHARING:
Plan to Share IPD: No